CLINICAL TRIAL: NCT00366106
Title: A Phase II, Open Label Study Evaluating an Alternative Schedule of Velcade/Dexamethasone Plus Doxil in the Treatment of Multiple Myeloma
Brief Title: Alternative Schedule of Velcade/Dexamethasone Plus Doxil for Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed to enrollment when it became clear that enrollment was too slow to complete full enrollment target within time frame allowed.
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACORN ALJBMM0502
Record Dates: First submitted 2006-08-16; First posted 2006-08-18 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bortezomib — Patients will be treated with bortezomib at 1.3mg/m^2 on Days 1, 4, 15, and 18 every 28 days (cycle).
  Other Names: Velcade
Drug: dexamethasone — Dexamethasone tablets will be given at 20mg daily on Days 1, 2, 4, 5, 15, 16, 18, and 19 every 28 days (cycle).
  Other Names: Decadron
Drug: doxorubicin HCl liposome — Patients will receive intravenous doxorubicin HCl liposome injection given at 30 mg/m^2 on Day 4 every 28 days (cycle).
  Other Names: Doxil

SUMMARY:
The current study is being conducted to evaluate the possibility that a different schedule of bortezomib, doxorubicin HCl liposome, and dexamethasone might decrease the incidence of peripheral neuropathy yet maintain similar efficacy and allow maintenance of bortezomib dosing for a longer period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient has confirmed diagnosis of relapsed/refractory multiple myeloma with measurable disease by serum or urine. Measurable disease defined as monoclonal protein of ≥ 1g/dl on serum protein electrophoresis (SPEP) or > 200 mg urine M protein/ 24 hours
* Patient has received at least 1 prior treatment regimen. (Prior treatment with bortezomib is allowed.)
* Patient has ECOG ≤ 2
* Patient provides voluntary written informed consent before performance of any study-relates procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Patients who have received prior high dose chemotherapy with stem cell support are eligible for this study.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

* Patient has a platelet count of < 50, 000 cells/mm³, within 14 days before enrollment.
* Patient has an absolute neutrophil count (ANC) ≤ 750/mm³ within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance of < 20 mL/min within 14 days before enrollment and/or serum creatinine ≥ 2.5 mg/dl.
* Patient has hemoglobin < 7.5 g/dl.
* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant.
* Patient has received a total cumulative dosage of anthracyclines exceeding 550 mg/m2.
* Patient has hypersensitivity to boron or mannitol.
* Patient has history of hypersensitivity reactions to a conventional formulation of doxorubicin HCl or the components of DOXIL.
* Patient has clinically significant coexisting illness unrelated to myeloma.
* Patient has uncontrolled diabetes.
* Patient has plasma cell leukemia.
* Patient has serum bilirubin > 1.5 x upper normal limit, alanine aminotransaminase (ALT), aspartate aminotransferase (AST) > 2.5 x upper normal limit (ULN), or alkaline phosphatase > 2.5 x ULN.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (B-hCG)pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs within 14 days before enrollment.
* Patient has serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnetta Blakely, MD, Principal Investigator — Accelerared Community Oncology Research Network, Inc.
Locations (15):
- United States (15):
  - Wilshire Oncology Medical Group, Inc., La Verne, California
  - Medical Oncology & Hematology, Waterbury, Connecticut
  - Advanced Medical Specialties, Miami, Florida
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Augusta Oncology Associates, PC, Augusta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Oncology-Hematology Associates, P.A., Clinton, Maryland
  - Hematology Oncology Centers of the Northern Rockies, PC, Billings, Montana
  - Arena Oncology Associates, Lake Success, New York
  - Tri-County Hematology and Oncology Associates, Canton, Ohio
  - Mid Ohio Oncology/Hematology, Inc., Columbus, Ohio
  - Lancaster Cancer Center, Ltd., Lancaster, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Cancer Specialists of Tidewater, Ltd., Chesapeake, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 community oncology research sites across the US within the ACORN network participated in this study. Enrollment started in July 2006 but was stopped in December 2008 at the point when it became clear that enrollment was too slow to complete the planned enrollment target of 45 patients within the time frame allowed.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent screening procedures to verify eligibility.
Groups:
- Treatment Group: All subjects received bortezomib 1.3mg/m^2 on Days 1, 4, 15, and 18 every 28 days and dexamethasone 20mg daily on Days 1, 2, 4, 5, 15, 16, 18, and 19 every 28 days. Following US FDA approval of doxorubicin HCl liposome injection in combination with bortezomib in May 2007, the study was amended to allow combination treatment with both bortezomib and doxorubicin HCl liposome injection 30 mg/m^2 on Day 4 every 28 days with dexamethasone. The target goal was 8 cycles of treatment.
Period: Overall Study
Arm/Group | Treatment Group
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 63.7 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Peripheral Neuropathy
Time Frame: Every 4 weeks from start of treatment until end of treatment
Measure: Number; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 32
Participants | 11

2. Secondary Outcome: Time to Progression (TTP)
Time Frame: TTP was measured from day 1 of treatment until time of progression, assessed up to 40 months
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Treatment Group
Number analyzed (Participants) | 32
Months | 23.07 (3.20)

3. Secondary Outcome: Number of Participants With Treatment Response
Description: Complete Response (CR), Partial Response (PR), and Minor Response (MR) each required stable bone disease and normal calcium levels. CR also required 100% serum protein electrophoresis (SPEP) reduction, negative immunofixation (IF), 100% urine protein electrophoresis (UPEP)reduction, and <5% plasma cells in bone marrow. PR also required >=50% SPEP reduction, >=90% UPEP reduction, and >=50% reduction in plasma cells in bone marrow. MR also required >=25% SPEP reduction, >=50% UPEP reduction, and > 25% reduction in plasma cells.
Time Frame: Every 8 weeks from start of treatment until end of treatment
Measure: Number; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 32
Participants | NA — We were unable to assess participant response to treatment due to missingness of data required for determination of response.

4. Secondary Outcome: Relative Dose Intensity of Bortezomib
Description: Relative dose intensity is defined as actual dose/scheduled dose. Bortezomib is administered on Days 1, 4, 15, and 18 every 28 days.
Time Frame: Each dose of bortezomib (days 1, 4, 15, and 18 every 28 days)
Population: Note that the sample sized varied at each dose and ranged from 32 patients to 1 patient.
Measure: Mean (Standard Deviation); unit: Relative dose intensity
Arm/Group | Treatment Group
Number analyzed (Participants) | 32
Relative dose intensity
  Cycle 1 / Week 1 | 0.97 (0.158)
  Cycle 1 / Week 1 Day 4 | 0.98 (0.159)
  Cycle 1 / Week 3 | 0.97 (0.158)
  Cycle 1 / Week 3 Day 18 | 0.97 (0.154)
  Cycle 2 / Week 5 | 0.95 (0.144)
  Cycle 2 / Week 5 Day 4 | 0.96 (0.148)
  Cycle 2 / Week 7 | 0.95 (0.140)
  Cycle 2 / Week 7 Day 18 | 0.96 (0.146)
  Cycle 3 / Week 9 | 0.99 (0.147)
  Cycle 3 / Week 9 Day 4 | 0.97 (0.121)
  Cycle 3 / Week 11 | 0.97 (0.142)
  Cycle 3 / Week 11 Day 18 | 0.95 (0.104)
  Cycle 4 / Week 13 | 0.99 (0.152)
  Cycle 4 / Week 13 Day 4 | 0.96 (0.111)
  Cycle 4 / Week 15 | 0.99 (0.154)
  Cycle 4 / Week 15 Day 18 | 0.96 (0.111)
  Cycle 5 / Week 17 | 0.98 (0.151)
  Cycle 5 / Week 17 Day 4 | 0.96 (0.110)
  Cycle 5 / Week 19 | 1.00 (0.157)
  Cycle 5 / Week 19 Day 18 | 0.97 (0.111)
  Cycle 6 / Week 21 | 1.01 (0.162)
  Cycle 6 / Week 21 Day 4 | 0.98 (0.114)
  Cycle 6 / Week 23 | 1.01 (0.169)
  Cycle 6 / Week 23 Day 18 | 0.99 (0.115)
  Cycle 7 / Week 25 | 1.11 (0.154)
  Cycle 7 / Week 25 Day 4 | 1.03 (0.148)
  Cycle 7 / Week 27 | 1.08 (0.198)
  Cycle 7 / Week 27 Day 18 | 1.03 (0.148)
  Cycle 8 / Week 29 | 1.05 (0.213)
  Cycle 8 / Week 29 Day 4 | 0.99 (0.140)
  Cycle 8 / Week 31 | 1.05 (0.213)
  Cycle 8 / Week 31 Day 18 | 1.04 (0.085)
  Cycle 9 / Week 33 | 1.10 (0.488)
  Cycle 9 / Week 33 Day 4 | 0.75 (NA) — Only 1 patient was dosed.
  Cycle 9 / Week 35 | 1.15 (0.417)
  Cycle 10 / Week 37 | 1.22 (0.311)
  Cycle 10 / Week 37 Day 4 | 1.00 (NA) — Only 1 patient was dosed.
  Cycle 10 / Week 39 | 1.22 (0.311)
  Cycle 10 / Week 39 Day 18 | 1.00 (NA) — Only 1 patient was dosed.
  Cycle 11 / Week 41 | 1.22 (0.311)
  Cycle 11 / Week 41 Day 4 | 1.00 (NA) — Only 1 patient was dosed.
  Cycle 11 / Week 43 | 1.44 (NA) — Only 1 patient was dosed.
  Cycle 11 / Week 43 Day 18 | 1.00 (NA) — Only 1 patient was dosed.

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning on day 1 of study treatment until one month after the end of study treatment.
Description: Systematic Assessment - subjects were assessed for adverse events weekly by either the research coordinator, treating physician, or other appropriate sub-investigator.
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 10/32
Other Adverse Events (participants affected / at risk) | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=32)
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Cellulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperglycemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=32)
Anemia (Blood and lymphatic system disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hemorrhagic diathesis (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Eye discharge (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Ocular surface disease (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Oral pain (Gastrointestinal disorders) | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
Chills (General disorders) | 1
Face edema (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 9
Lethargy (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Edema peripheral (General disorders) | 7
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Abscess jaw (Infections and infestations) | 1
Adenoviral upper respiratory infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 4
Oral fungal infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infections (Infections and infestations) | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Barotitis media (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Vaginal laceration (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatine increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood potassium increased (Investigations) | 3
Blood urea decreased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 1
Hemoglobin decreased (Investigations) | 2
Heart rate increased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Amnesia (Nervous system disorders) | 1
Burning feet syndrome (Nervous system disorders) | 1
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Hypoesthesia (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 11
Paresthesia (Nervous system disorders) | 5
Parosmia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 4
Nervousness (Psychiatric disorders) | 1
Renal tubular acidosis (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vaginal mucosal blistering (Reproductive system and breast disorders) | 1
Vulvovaginal pruritis (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Skin discoloration (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Ecchymosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was closed to enrollment when it became clear that enrollment was too slow to complete the planned enrollment target of 45 patients within the time frame allowed. Response rate was unable to be assessed due to missingness of required data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the disclosure must be given to Millennium for review at least 30 days before it is submitted for publication or disclosure. If a Development is contained in the disclosure, Research Organization and/or Principal Investigator defer publication or disclosure for 90 days from the time Millennium notifies that it wants to file a patent application on the Development provided such notice was provided by Millennium within 30 days of the copy first provided to Millennium.